CLINICAL TRIAL: NCT03744676
Title: A Safety Trial of Lisocabtagene Maraleucel (JCAR017) for Relapsed and Refractory (R/R) B-cell Non-Hodgkin Lymphoma (NHL) in the Outpatient Setting
Brief Title: A Safety Trial of Lisocabtagene Maraleucel (JCAR017) for Relapsed and Refractory (R/R) B-cell Non-Hodgkin Lymphoma (NHL) in the Outpatient Setting (TRANSCEND-OUTREACH-007)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Juno Therapeutics, a Subsidiary of Celgene (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 017007
Record Dates: First submitted 2018-11-07; First posted 2018-11-16 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Neoplasms; Neoplasms by Histologic Type; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Disorder
Keywords: Lisocabtagene maraleucel; liso-cel; JCAR017; relapse; refractory; B-Cell Non-Hodgkin Lymphoma; NHL; chimeric antigen receptor; CAR; CAR T cell; autologous T cell therapy; immunotherapy; cell therapy; B-cell malignancies
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Neoplasms; Neoplasms by Histologic Type; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lisocabtagene maraleucel (Experimental): Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of lisocabtagene maraleucel. During lisocabtagene maraleucel production, subjects may receive low-dose chemotherapy for disease control. Upon successful generation of lisocabtagene maraleucel product, subjects will receive treatment which will include lymphodepleting chemotherapy followed by one dose of lisocabtagene maraleucel administered by intravenous (IV) injection.
  Interventions: Biological: lisocabtagene maraleucel

INTERVENTIONS:
Biological: lisocabtagene maraleucel — lisocabtagene maraleucel will be administered as single dose intravenous (IV) injection
  Other Names: JCAR017; liso-cel

SUMMARY:
This is an open-label, multicenter, Phase 2 study to determine the safety, PK, and efficacy of lisocabtagene maraleucel (JCAR017) in subjects who have relapsed from, or are refractory to, two lines of immunochemotherapy for aggressive B-cell non-Hodgkin lymphoma (NHL) in the outpatient setting. Subjects will receive treatment with JCAR017 and will be followed for up to 2 years.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 2 study to assess the safety and antitumor activity in adult patients with relapsed or refractory B-cell non-Hodgkin Lymphoma when administered with lisocabtagene maraleucel (JCAR017) in the outpatient setting.

Upon the successful product generation of lisocabtagene maraleucel, subjects will enter the treatment phase of the study. Treatment will include lymphodepleting chemotherapy followed by lisocabtagene maraleucel administration. Subjects will then enter the post-treatment follow-up phase of the study and will be followed for approximately 24 months for safety, disease status, health-related quality of life (HRQoL), and survival. Long-term follow-up will continue under a separate long-term follow-up protocol, per health regulatory authority guidelines, currently up to 15 years after the last lisocabtagene maraleucel administration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of consent
* Relapsed or refractory B-cell NHL of the following histologies: diffuse large B cell lymphoma (DLBCL) not otherwise specified; includes biopsy-confirmed transformed DLBCL from indolent histologies, high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements with DLBCL histology, primary mediastinal B-cell lymphoma(PMBCL), and follicular lymphoma Grade 3B. Subjects must have been treated with an anthracycline and rituximab (or other CD20-targeted agent) and have relapsed or refractory disease after at least 2 systemic lines of therapy for DLBCL or after auto-HSCT.
* Positron-emission tomography-positive disease by Lugano Classification
* Eastern Cooperative Oncology Group performance status of 0 to 1
* Adequate bone marrow, renal, hepatic, pulmonary, cardiac organ function
* Adequate vascular access for leukapheresis procedure
* Subjects who have received previous CD19-targeted therapy must have CD19-positive lymphoma confirmed on a biopsy since completing the prior CD19-targeted therapy
* Subjects must agree to use appropriate contraception.

Exclusion Criteria:

* Subjects with central nervous system (CNS)-only involvement by malignancy (note: subjects with secondary CNS involvement are allowed on study)
* History of prior allogeneic hematopoietic stem cell transplant
* Treatment with alemtuzumab within 6 months of leukapheresis, or treatment with fludarabine or cladribine within 3 months of leukapheresis
* History of another primary malignancy that has not been in remission for at least 2 years.The following are examples of exceptions from the 2-year limit: nonmelanoma skin cancer, definitively-treated stage 1 solid tumor with a low risk of recurrence, curatively treated localized prostate cancer, and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on a Papanicolau smear.
* Active hepatitis B or hepatitis C infection at the time of screening
* History of or active human immunodeficiency virus infection at the time of screening
* Uncontrolled systemic fungal, bacterial, viral or other infection despite appropriate anti-infection treatment at the time of leukapheresis or lisocabtagene maraleucel administration
* Presence of acute or chronic graft-versus-host disease
* History of clinically significant cardiac conditions within the past 6 months
* History or presence of clinically relevant CNS pathology such as epilepsy/seizure, paresis, aphasia, stroke, cerebral edema, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
* Pregnant or nursing women
* Subject does not meet protocol-specified washout periods for certain prior treatments
* Prior CAR T-cell or other genetically modified T-cell therapy
* Progressive vascular tumor invasion, thrombosis, or embolism
* Venous thrombosis or embolism not managed on stable regimen of anticoagulation
* Uncontrolled medical, psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (23):
- United States (23):
  - Local Institution - 0057, Los Angeles, California
  - Local Institution - 0060, Denver, Colorado
  - Local Institution - 0089, Miami, Florida
  - Local Institution - 0081, Orlando, Florida
  - Local Institution - 0065, Indianapolis, Indiana
  - Local Institution - 0069, Wichita, Kansas
  - Local Institution - 0064, Louisville, Kentucky
  - Local Institution - 0101, Southfield, Michigan
  - Local Institution - 0052, East Brunswick, New Jersey
  - Local Institution - 0066, Morristown, New Jersey
  - Local Institution - 0041, Albany, New York
  - Local Institution - 0039, Cincinnati, Ohio
  - Local Institution - 0098, Eugene, Oregon
  - Local Institution - 0051, Portland, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Local Institution - 0037, Greenville, South Carolina
  - Local Institution - 0063, Nashville, Tennessee
  - Local Institution - 0097, Dallas, Texas
  - Local Institution - 0061, San Antonio, Texas
  - Baylor Scott and White Health, Temple, Texas
  - Local Institution - 0096, Tyler, Texas
  - Local Institution - 0074, Salt Lake City, Utah
  - Local Institution - 0036, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- [Derived] Linhares Y, Freytes CO, Cherry M, Bachier C, Maris M, Hoda D, Varela JC, Bellomo C, Cross S, Essell J, Fanning S, Terebelo H, Yimer H, Courtright J, Sharman JP, Kostic A, Vedal M, Ogasawara K, Avilion A, Espinola R, Yuan B, Mattar B. OUTREACH: phase 2 study of lisocabtagene maraleucel as outpatient or inpatient treatment at community sites for R/R LBCL. Blood Adv. 2024 Dec 10;8(23):6114-6126. doi: 10.1182/bloodadvances.2024013254. PMID 39347584
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Groups:
- Lisocabtagene Maraleucel (JCAR017): Participants underwent leukapheresis and may receive salvage low- dose chemotherapy or one cycle of non-curative standard of care antitumor therapy if required. Eligible participants then received lymphodepleting chemotherapy with fludarabine and cyclophosphamide (flu/cy) followed by a single dose of JCAR017 (100×10^6 CAR+ T cells/infusion) administered intravenously (IV) 2 to 7 days after completion of lymphodepleting chemotherapy.
Period: Pre-Treatment Phase
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Started (Participants who underwent leukapheresis) | 104
Completed (Participants who completed leukapheresis and continued to lymphodepleting chemotherapy (LDC) treatment period and JCAR017) | 84
Not Completed | 20
Not completed — Disease related complications | 2
Not completed — No longer meets study criteria | 4
Not completed — Death | 7
Not completed — Other Reasons | 7
Period: Treatment Phase
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Started (Participants who underwent lymphodepleting chemotherapy (LDC) treatment with conforming JCAR017) | 82
Participants Who Received LDC and Non Conforming Product | 1
Completed (Completed study) | 35
Not Completed | 47
Not completed — Participant withdrew consent | 8
Not completed — Death | 33
Not completed — other reasons | 6

BASELINE CHARACTERISTICS:
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 104
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.9 (11.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 77
  Unknown or Not Reported | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 88
    Other | 7
    Unknown | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Cytokine Release Syndrome (CRS) Adverse Events Grade ≥ 3
Description: Cytokine release syndrome is characterized by high fever, fatigue, nausea, headache, dyspnea, tachycardia, rigors, hypotension, hypoxia, myalgia/arthralgia, and anorexia.
  Incidence of Grade ≥ 3 CRS, based on the TEAE with MedDRA PT "Cytokine release syndrome," graded according to the grading scale adapted from Lee (Lee 2014).
Time Frame: From first dose to 90 days following first dose (up to approximately 90 days)
Population: All participants who received at least one JCAR017 infusion
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Percentage of participants | 0.0 [0.0 to 4.4]

2. Primary Outcome: Percentage of Participants With Neurotoxicity (NT) Adverse Events Grade ≥ 3
Description: NT events have also been reported and may include neurologic symptoms such as altered mental status, aphasia, altered level of consciousness, and seizures or seizure-like activity.
  Incidence of Grade ≥ 3 NT, defined as an Investigator-identified TEAE considered neurotoxicity related to JCAR017.
Time Frame: From first dose to 90 days following first dose (up to approximately 90 days)
Population: All participants who received at least one JCAR017 infusion
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Percentage of participants | 9.8 [4.3 to 18.3]

3. Primary Outcome: Percentage of Participants With Infection Adverse Events Grade ≥ 3
Description: Incidence of treatment-emergent Grade ≥ 3 infections, defined using MedDRA SOC.
Time Frame: From first dose to 90 days following first dose (up to approximately 90 days)
Population: All participants who received at least one JCAR017 infusion
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Percentage of participants | 11.0 [5.1 to 19.8]

4. Primary Outcome: Percentage of Participants With Grade ≥ 3 Prolonged Cytopenia at Day 29.
Description: Prolonged cytopenia is defined as the occurrence of Grade ≥ 3 cytopenia not resolved by the Day 29 visit, based on laboratory results of low hemoglobin, absolute neutrophil count decreased, and platelet count decreased. The frequency of subjects experiencing each individual laboratory abnormality and the total number with at least 1 abnormality will be summarized, as will recovery from prolonged cytopenia after Day 29.
Time Frame: At Day 29 after first treatment
Population: All participants who received at least one JCAR017 infusion
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Percentage of participants | 32.9 [22.9 to 44.2]

5. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: From first dose to 90 days following first dose (up to approximately 90 days)
Population: All participants who received at least one JCAR017 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Participants | 82

6. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities- Hematology
Time Frame: From first dose to up to 41 months
Population: All participants who received at least one JCAR017 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Participants | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities- Chemistry
Time Frame: From first dose to up to 41 months
Population: All participants who received at least one JCAR017 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Participants | 0

8. Secondary Outcome: Number of Participants With Adverse Events Grade ≥ 3
Time Frame: From first dose to 90 days following first dose (up to approximately 90 days)
Population: All participants who received at least one JCAR017 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Participants | 61

9. Secondary Outcome: Time to Onset and Time to Resolution of Grade ≥ 3 Cytokine Release Syndrome (CRS)
Time Frame: From first dose to up to approximately 41 months
Population: All participants who received at least one JCAR017 infusion
Measure: Median (Full Range); unit: Days
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Days
  Time to Onset | 0 [0 to 0]
  Time to Resolution | 0 [0 to 0]

10. Secondary Outcome: Time to Onset and Time to Resolution of Grade ≥ 3 Neurotoxicity (NT)
Time Frame: From first dose to up to approximately 41 months
Population: All participants who received at least one JCAR017 infusion
Measure: Median (Full Range); unit: Days
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Days
  Time to Onset: number analyzed (Participants) | 8
  Time to Onset | 9.5 [3 to 33]
  Time to Resolution: number analyzed (Participants) | 8
  Time to Resolution | 16.5 [5 to 47]

11. Secondary Outcome: Number of Participants Administered Tocilizumab and Corticosteroid for Management of Cytokine Release Syndrome (CRS)
Time Frame: From first dose to up to approximately 41 months
Population: All participants who received at least one JCAR017 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Participants
  Tocilizumab Only | 7
  Corticosteroid Only | 2
  Both Tocilizumab and Corticosteroid | 7

12. Secondary Outcome: Number of Participants Administered Tocilizumab and Corticosteroid for Management of Neurotoxicity (NT)
Time Frame: From first dose to up to study completion (Approximately 57 Months and 24 days)
Population: All participants who received at least one JCAR017 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Participants
  Tocilizumab Only | 0
  Corticosteroid Only | 12
  Both Tocilizumab and Corticosteroid | 1

13. Secondary Outcome: Objective Response Rate (ORR)
Description: The Percentage of participants with a best overall response (BOR) of either CR or PR based on the Lugano 2014 criteria.
  Disease response will be determined according to the "Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification"
  Complete response is defined as:
  1. Score 1, 2, or 3a with or without residual mass
  2. No evidence of FDG-avid disease in marrow
  Partial Response is defined as:
  1. Score 4 or 5a with reduced uptake compared with baseline and residual masses of any size
  2. Bone marrow with residual uptake higher than in normal marrow but reduced compared with baseline (diffuse uptake compatible with reactive changes from chemotherapy allowed). If there are persistent focal changes in marrow in the context of a nodal response, should consider further evaluation with MRI, biopsy, or interval scan.
Time Frame: From first dose to up to approximately 41 months
Population: All participants who received at least one JCAR017 infusion
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Percentage of Participants | 80.5 [70.3 to 88.4]

14. Secondary Outcome: Complete Response Rate (CRR)
Description: The Percentage of participants with a best overall response (BOR) with CR based on the Lugano 2014 criteria.
  Disease response will be determined according to the "Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification"
  Complete response is defined as:
  1. Score 1, 2, or 3a with or without residual mass
  2. No evidence of FDG-avid disease in marrow
Time Frame: From first dose to up to approximately 41 months
Population: All participants who received at least one JCAR017 infusion
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Percentage of Participants | 53.7 [42.3 to 64.7]

15. Secondary Outcome: Duration of Response (DoR) and Duration of Complete Response (DoCR)
Description: Duration of response (DOR) is defined as the time from the first documentation of response (CR or PR) after JCAR017 infusion to disease progression or death from any cause, whichever occurs first.
  Duration of response (DOR) if BOR is CR is defined for subjects with a BOR of CR as the time from the first documentation of response (CR or PR) after JCAR017 infusion to earlier of disease progression or death from any cause.
Time Frame: From first dose to up to approximately 41 months
Population: All participants who received at least one JCAR017 infusion
Measure: Median (Full Range); unit: Months
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Months
  DoR | 14.75 [5.03 to NA] — Insufficient number of participants with a response to reach upper limit number according to KM methodology.
  DoCR: number analyzed (Participants) | 44
  DoCR | NA [16.59 to NA] — Insufficient number of participants with a response to reach median upper limit number according to KM methodology.

16. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival is defined as the time from infusion of JCAR017 to progressive disease or death, whichever is earlier. If a subject does not have an event for the PFS analysis, the subject will be censored.
  Progressive Disease is defined as:
  1. Score 4 or 5a with an increase in intensity of uptake from nadir
  2. New FDG-avid foci consistent with lymphoma (may need biopsy or repeat scan if uncertain about etiology of foci).
  3. Investigator assessed clinical progression
Time Frame: From first dose to up to study completion (Approximately 57 Months and 24 days)
Population: All participants who received at least one JCAR017 infusion
Measure: Median (Full Range); unit: Months
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Months | 5.86 [0.7 to 26.7]

17. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from infusion of JCAR017 to the date of death. For assessment of OS, data from surviving participants will be censored at the last time that the participant is known to be alive. The OS analysis will include all available survival information from the long-term follow-up study if applicable.
Time Frame: From first dose to up to study completion (Approximately 57 Months and 24 days)
Population: All participants who received at least one JCAR017 infusion
Measure: Median (Full Range); unit: Months
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Months | 21.88 [1.0 to 50.1]

18. Secondary Outcome: Area Under the Blood Concentration-time Curve From Time to Zero to 28 Days After Dosing AUC (0-28)
Time Frame: 28days after first dose
Population: qPCR PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*copies/μg
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 81
day*copies/μg | 219760.3 (216.1)

19. Secondary Outcome: Maximum Observed Blood Concentration (Cmax)
Time Frame: 28days after first dose
Population: qPCR PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/μg
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 81
copies/μg | 24077.8 (230.7)

20. Secondary Outcome: Time of Maximum Observed Blood Concentration (Tmax)
Time Frame: 28days after first dose
Population: qPCR PK Analysis Set
Measure: Median (Full Range); unit: days
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 81
days | 10.0 [7 to 28]

21. Secondary Outcome: Mean Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30
Description: The EORTC QLQ-C30 is a 30-item scale composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A higher scale score represents a higher level of well-being and better ability of daily functioning. Thus, a high score for a functional scale represents a high/healthy level of functioning; a high score for the global health status/HRQoL represents a high HRQoL, but a high score for a symptom scale/item represents a high level of symptomatic problem.
Time Frame: From Enrollment to end of follow up, approximately 26 months
Population: JCAR017 All treated participants with a measurement at post dose month 24
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 22
Scores on a Scale
  Apptetie Loss | -22.7 (23.87)
  Cognitive Functioning | 1.5 (18.48)
  Constipation | -7.6 (27.08)
  Diarrhea | -3.0 (27.04)
  Dyspnea | 6.1 (13.16)
  Emotional Functioning | 2.7 (20.31)
  Fatigue | -14.6 (21.24)
  Financial Difficulties | -9.1 (25.58)
  Global Health Stuats/QoL | 15.2 (21.61)
  Insomnia | -10.6 (27.96)
  Nausea and Vomiting | -9.8 (17.56)
  Pain | -13.6 (26.55)
  Physical Functioning | 2.4 (16.14)
  Role Functioning | 12.9 (23.53)
  Social Functioning | 17.4 (24.92)

22. Secondary Outcome: Mean Change From Baseline in EuroQol Instrument EQ-5D-5L.
Description: The European Quality of Life 5D-5L Scale (EQ-5D-5L) assesses general health-related quality of life. Health is defined in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded so that a '1' indicates no problem, and '5' indicates the most serious problem. The responses for the 5 dimensions are combined in a 5-digit number. The EQ-5D-5L health utility index (HUI) is assessed using the Crosswalk algorithm for France based on the individual responses to the 5 EQ-5D-5L domains ranging from -0.530 to 1.000. The smallest change considered clinically meaningful, is defined as a score difference of 0.08 points.
Time Frame: Post Dose Month 24
Population: All treated participants with an EQ-5D-5L index score post dose month 24
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 21
Score on a Scale | 0.0 (0.13)

23. Secondary Outcome: Number of Intensive Care Unit (ICU) Inpatient Days and Non-ICU Inpatient Days and Reasons for Hospitalization
Description: Length of initial ICU and non-ICU stay from liso-cel administration
Time Frame: From first hospitalization to the last. Approximately 31 days
Population: Liso-cel-treated Analysis Set - Inpatient Monitored
Measure: Median (Full Range); unit: days
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 25
days
  Initial ICU Stay: number analyzed (Participants) | 2
  Initial ICU Stay | 5.5 [4 to 7]
  Initial Non-ICU Stay | 15.0 [0 to 31]

24. Secondary Outcome: Number of Participants Who Received Transfusions
Description: Number of participants who received transfusions
Time Frame: From first dose to end of treatment period approximately 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Participants | 43

25. Secondary Outcome: Number of Participants Requiring Growth Factor Support.
Description: Growth factor support was defined as concomitant administration of FILGRASTIM, TBO FILGRASTIM, PEGFILGRASTIM, FILGRASTIM SNDZ, or FILGRASTIM AAFI.
Time Frame: From first dose to end of treatment period approximately 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Participants | 35

26. Secondary Outcome: Number of Participants Requiring Intravenous Immunoglobulin (IVIG) Support
Description: Number of participants requiring intravenous immunoglobulin (IVIG) support
Time Frame: From first dose to end of treatment period approximately 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
Number analyzed (Participants) | 82
Participants | 12

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose until study completion (up to approximately 57 months and 24 days). SAEs and Other AEs were assessed from first dose to 90 days following first dose (up to approximately 90 days).
Description: The total number at risk for all-cause mortality represents all participants who underwent leukapheresis. The total number at risk by any serious adverse event and other (not including serious) adverse events represents all participants that received at least 1 dose of study medication (JCAR017).
Arm/Group | Lisocabtagene Maraleucel (JCAR017)
All-Cause Mortality (participants affected / at risk) | 48/82
Serious Adverse Events (participants affected / at risk) | 48/82
Other Adverse Events (participants affected / at risk) | 82/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lisocabtagene Maraleucel (JCAR017) (N=82)
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Gait disturbance (General disorders) | 1
Pyrexia (General disorders) | 4
Cytokine release syndrome (Immune system disorders) | 24
Atypical pneumonia (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 2
Clostridium difficile colitis (Infections and infestations) | 1
Cytomegalovirus viraemia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 4
Demyelinating polyneuropathy (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Memory impairment (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Slow speech (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 4
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 2
Delirium (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Hallucination, visual (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lisocabtagene Maraleucel (JCAR017) (N=82)
Anaemia (Blood and lymphatic system disorders) | 28
Leukopenia (Blood and lymphatic system disorders) | 36
Lymphopenia (Blood and lymphatic system disorders) | 17
Neutropenia (Blood and lymphatic system disorders) | 55
Thrombocytopenia (Blood and lymphatic system disorders) | 29
Abdominal pain (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 19
Diarrhoea (Gastrointestinal disorders) | 19
Nausea (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 8
Asthenia (General disorders) | 9
Fatigue (General disorders) | 25
Oedema peripheral (General disorders) | 10
Pyrexia (General disorders) | 12
Cytokine release syndrome (Immune system disorders) | 10
Hypogammaglobulinaemia (Immune system disorders) | 7
Fall (Injury, poisoning and procedural complications) | 5
Decreased appetite (Metabolism and nutrition disorders) | 19
Dehydration (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 20
Lethargy (Nervous system disorders) | 6
Tremor (Nervous system disorders) | 8
Agitation (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 7
Hypotension (Vascular disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT03744676/Prot_SAP_000.pdf